CLINICAL TRIAL: NCT03346980
Title: Endoscopic Evaluation of Duodenal Polyposis in Patients With Familial Adenomatous Polyposis (FAP) - a Single Center Prospective Validation of the Spigelman Classification
Brief Title: Endoscopic Evaluation of Duodenal Polyposis in Patients With Familial Adenomatous Polyposis (FAP)
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, John Gasdal Karstensen, Principal Investigator, Copenhagen University Hospital, Hvidovre
Other Study IDs: SPIGELMAN-VALIDATE
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Familial Adenomatous Polyposes; Duodenal Polyposis; Duodenal Cancer
Keywords: Spigelman
MeSH Terms: conditions — Adenomatous Polyposis Coli; Duodenal Neoplasms | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Familial adenomatous polyposis: The Danish Polyposis Register is sited at Copenhagen University Hospital Hvidovre. From this registry consecutive familial adenomatous polyposis patients referred for esophagogastroduodenoscopy (EGD) will prospectively be enrolled in this single-center study. Both patients referred for endoscopic surveillance and interventional endoscopy are eligible.
  Interventions: Diagnostic Test: Esophagogastroduodenoscopy

INTERVENTIONS:
Diagnostic Test: Esophagogastroduodenoscopy — All patients will be evaluated with both standard HD gastroscope and side-viewing duodenoscope; the latter to ensure proper visualization of the major papilla.

SUMMARY:
Familial adenomatous polyposis (FAP) is an autosomal dominant genetic disorder that predisposes to a number or malignant disorders [1,2]. Clinically, FAP presents with an abnormal number of colorectal polyps (100-5000), while it genetically is defined by mutations in the APC-gene [1]. Historically, colorectal cancer has been the major cause of deaths for FAP patient. However, as the incidence of colorectal cancer has decreased with the use of prophylactic colectomy, the incidence of duodenal cancer has increased [3,4]. It is estimated that the cumulative lifetime risk of duodenal polyposis exceeds 95% [1,5]. The predictor of duodenal cancer is duodenal polyposis, which is almost inevitable in patients with FAP.

In 1989 the Spigelman score was introduced in order to assess the severity of duodenal polyposis and stratify patients according to risk of duodenal cancer (Table 1) [6]. It is a composite score that includes two endoscopic parameters (number and maximum size of polyps, respectively) and two histopathological parameters (histological subtype and grade of dysplasia). The score ranges from 0-12 and it has been classified in four stages. The 10-year risk of developing duodenal cancer corresponds with the Spigelman stage ranging from ≈0 for stage 0-1 to 36% for stage 4 [7]. Besides duodenal cancer, the indications of cancer prophylactic surgical resection are debatable, but generally recommended in the case of Spigelman stage 4 or high-grade dysplasia.

Table 1 Spigelman Classification for duodenal polyposis Criterion 1 point 2 points 3 points Polyp number 1-4 5-20 >20 Polyp size (mm) 1-4 5-10 >20 Histology Tubular Tubulovillous Villous Dysplasia Low grade* High grade* Stage 0: 0 points; stage I: 1-4 points; stage II: 5-6 points; stage III: 7-8 points; stage IV: 9-12 points. *Originally, 3 grades of dysplasia were incorporated.

While the correlation to cancer has been explored in several studies, the validation and the reproducibility of the Spigelman score remains somewhat unclear. The primary aim of this study is to assess the inter- and intra-observer agreement of the Spigelman score for experienced endoscopists using state-of-the-art high-definition (HD) endoscopes.

Hypothesis: The Spigelman score has perfect reproducibility for endoscopic experts (κ>0.80 with 95% CI.).

DETAILED DESCRIPTION:
The Danish Polyposis Register is sited at Copenhagen University Hospital Hvidovre. From this registry consecutive FAP patients referred for esophagogastroduodenoscopy (EGD) will prospectively be enrolled in this single-center study. Both patients referred for endoscopic surveillance and interventional endoscopy are eligible.

All patients will be evaluated with both standard HD gastroscope and side-viewing duodenoscope; the latter to ensure proper visualization of the major papilla. Movie sequences will be saved for post-procedural evaluation. Any sedation or buscopan administered will be registered. A biopsy protocol according to the attached CRF will be followed carefully and furthermore, if any interventional procedures are carried out, they will be registered as well as the presence of any gastric adenomas. In general, the approach is considered standard care and the study does not differ from the treatment algorithm and the national guidelines.

Post-procedural, the movies will be evaluated by three expert endoscopists all having long-term experience with FAP patients. In order to assess the inter-observer agreement of the Spigelman score, the endoscopic sub-scores by the three experts will be combined with the histopathological data. Furthermore, the inter-observer agreement of the endoscopic sub-scores will be analyzed separately. To assess the intra-observer agreement, after a minimum of one week one of the expert endoscopists will undertake a second evaluation of the movies after they have been randomized. The precise same methodology will be carried out for three novices. All clinical details will be erased from the movies before evaluation.

Design: A blinded single-center prospective observation and methodology study with subsequent calculation of intra-and inter-observer variability.

Statistical method: Intra-and inter-observer agreements between 3 operators at for the Spigelman score are calculated by weighted kappa statistics (inter class correlation).

Patients: A complete sample-size calculation has been made for the inter-observer study of the 3 observers for the Spigelman Score. To estimate an expected ICC of 0.9 being significantly higher than a threshold at 0.8 with power of 0.8 and a one-sided significance level of 0.05, 33 patients need to be enrolled in the study per protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients known with FAP (having either an APC mutation, or >100 colorectal adenomas and a positive family history) and with an indication of EGD as part of their surveillance or therapeutic program.

Exclusion Criteria:

* Patients, in whom the standard biopsy protocol cannot be fulfilled due to vital anticoagulant therapy, liver failure etc.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Danish Polyposis Register is sited at Copenhagen University Hospital Hvidovre. From this registry consecutive FAP patients referred for esophagogastroduodenoscopy (EGD) will prospectively be enrolled in this single-center study. Both patients referred for endoscopic surveillance and interventional endoscopy are eligible.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Inter-observer agreement of the Spigelman Score evaluated by expert endoscopists. | 1 week
  The score ranges from 0-12 and it has been classified in four stages. The 10-year risk of developing duodenal cancer corresponds with the Spigelman stage ranging from ≈0 for stage 0-1 to 36% for stage 4. Stage 0: 0 points; stage I: 1-4 points; stage II: 5-6 points; stage III: 7-8 points; stage IV: 9-12 points.

SECONDARY OUTCOMES:
Inter- and intra-observer agreement of the endoscopic sub-scores evaluated by expert endoscopists (the number of polyps and the size of these) | 1 week
  The endoscopic subscores (the number of polyps and the size of these) will be analyzed separately.
Intra-observer agreement of Spigelman Score evaluated by expert endoscopists. | 1 week
  The score ranges from 0-12 and it has been classified in four stages. The 10-year risk of developing duodenal cancer corresponds with the Spigelman stage ranging from ≈0 for stage 0-1 to 36% for stage 4. Stage 0: 0 points; stage I: 1-4 points; stage II: 5-6 points; stage III: 7-8 points; stage IV: 9-12 points.
Inter- and intra-observer agreement of the Spigelman Score and the endoscopic sub-scores evaluated by novices. | 1 week
  The score ranges from 0-12 and it has been classified in four stages. The 10-year risk of developing duodenal cancer corresponds with the Spigelman stage ranging from ≈0 for stage 0-1 to 36% for stage 4. Stage 0: 0 points; stage I: 1-4 points; stage II: 5-6 points; stage III: 7-8 points; stage IV: 9-12 points. The endoscopic subscores (the number of polyps and the size of these) will be analyzed separately.

CONTACTS AND LOCATIONS:
Overall Officials: John G Karstensen, Principal Investigator — MD, PhD
Locations (1):
- Copenhagen University Hospital Hvidovre, Hvidovre, Capital, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vasen HF, Moslein G, Alonso A, Aretz S, Bernstein I, Bertario L, Blanco I, Bulow S, Burn J, Capella G, Colas C, Engel C, Frayling I, Friedl W, Hes FJ, Hodgson S, Jarvinen H, Mecklin JP, Moller P, Myrhoi T, Nagengast FM, Parc Y, Phillips R, Clark SK, de Leon MP, Renkonen-Sinisalo L, Sampson JR, Stormorken A, Tejpar S, Thomas HJ, Wijnen J. Guidelines for the clinical management of familial adenomatous polyposis (FAP). Gut. 2008 May;57(5):704-13. doi: 10.1136/gut.2007.136127. Epub 2008 Jan 14. PMID 18194984
- [Background] Bulow S, Bjork J, Christensen IJ, Fausa O, Jarvinen H, Moesgaard F, Vasen HF; DAF Study Group. Duodenal adenomatosis in familial adenomatous polyposis. Gut. 2004 Mar;53(3):381-6. doi: 10.1136/gut.2003.027771. PMID 14960520
- [Background] Spigelman AD, Williams CB, Talbot IC, Domizio P, Phillips RK. Upper gastrointestinal cancer in patients with familial adenomatous polyposis. Lancet. 1989 Sep 30;2(8666):783-5. doi: 10.1016/s0140-6736(89)90840-4. PMID 2571019